CLINICAL TRIAL: NCT00760578
Title: A Phase 2A, Randomized, Double-Blind, Comparator- and Placebo-Controlled, Multiple-Dose Study to Evaluate the Safety, Tolerability and Efficacy of Two Dose Levels of Mitoglitazone™ in Type 2 Diabetic Patients
Brief Title: A Placebo Controlled Safety and Efficacy Study of MSDC-0160 in Type 2 Diabetes With Active Comparator
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metabolic Solutions Development Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSDC-C003
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; MSDC-0160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Microcrystaline cellulose once daily
  Interventions: Drug: Placebo
- Pioglitazone (Active Comparator): Pioglitazone 45 mg once daily
  Interventions: Drug: Pioglitazone
- MSDC-0160 90 mg (Experimental): MSDC-0160 90 mg once daily
  Interventions: Drug: MSDC-0160 90 mg
- MSDC-0160 220 mg (Experimental): MSDC-0160 220 mg once daily
  Interventions: Drug: MSDC-0160 220 mg

INTERVENTIONS:
Drug: Placebo — Once daily, oral
  Arms: Placebo
Drug: Pioglitazone — Once daily, oral
  Arms: Pioglitazone
Drug: MSDC-0160 90 mg — Once daily, oral
  Arms: MSDC-0160 90 mg
Drug: MSDC-0160 220 mg — Once daily, oral
  Arms: MSDC-0160 220 mg

SUMMARY:
The purpose of this study is to determine if MSDC-0160 is effective in the treatment of Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes naive or on metformin
* Male and female (postmenopausal or surgically sterilized), 18 to 70 years of age.

Exclusion Criteria:

* Use of diabetes medications other than metformin.
* History of heart failure or previous myocardial infarction.
* Blood pressure great than 160/100 mmHg.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Colca, PhD, Study Director — Metabolic Solutions Development Company
Locations (8):
- United States (8):
  - Los Angeles, California
  - Miami Gardens, Florida
  - West Palm Beach, Florida
  - Kalamazoo, Michigan
  - Greenville, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Renton, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the United States by 10 investigators between 26 Sep 2008 and 02 Feb 2009.
Pre-assignment Details: This was a Ph 2A, double-blind, randomized, comparator- & placebo-controlled study of Mitoglitazone in otherwise healthy adult patients with type 2 diabetes. The study consisted of a maximum 21-day screening period, a 2 week, single-blind, placebo lead-in period, a 4 week, double-blind treatment period and a 1 week posttreatment follow-up period.
Period: Overall Study
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo
Started | 22 | 21 | 21 | 22
Entered Drug Treatment Period | 21 | 20 | 19 | 22
Completed | 19 | 19 | 16 | 18
Not Completed | 3 | 2 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 22 | 21 | 21 | 22 | 86
Age Continuous [Mean (Standard Deviation); unit: years] | 56.3 (8.20) | 53.7 (9.22) | 57.7 (6.38) | 54.5 (8.79) | 55.5 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 14 | 13 | 46
  Male | 12 | 12 | 7 | 9 | 40
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 21 | 22 | 86

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Averaged Postprandial Glucose in Response to a MMT Test
Description: Change from baseline of averaged postprandial glucose (mmol/L) in response to a Mixed-meal tolerance (MMT) test.
Time Frame: 28 days
Population: All patients who were compliant during the treatment period and who had a Day 8 and Day 43 averaged mixed-meal tolerance test and laboratory assessments. Compliance during the treatment period was determined by the sponsor through a manual review of pill counts, including a review of comments from the study sites.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- Mitoglitazone 90 mg: Mitoglitazone 90 mg taken once daily for 28 days
- Mitoglitazone 220 mg: Mitaglitazone 220 mg taken once daily for 28 days
- Pioglitazone 45 mg: Pioglitazone 45 mg taken once daily for 28 days
- Placebo: Placebo (microcrystalline cellulose) taken once daily for 28 days
Arm/Group | Mitoglitazone 90 mg | Mitoglitazone 220 mg | Pioglitazone 45 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
mmol/L | 0.16 (0.349) | -0.44 (0.358) | -1.10 (0.390) | 0.51 (0.340)

2. Secondary Outcome: Change From Baseline in Averaged Insulin Levels in Response to a Mixed-meal Tolerance Test
Description: Change from baseline in averaged post prandial insulin levels in response to a mixed-meal tolerance test.
Time Frame: After four weeks of active therapy
Population: All patients who were compliant during the treatment period and who had a Day 8 and Day 43 averaged mixed-meal tolerance (MMT) test and laboratory assessments. Compliance during the treatment period was determined by the sponsor through a manual review of pill counts, including a review of comments from the study sites.
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Groups:
- Placebo: Microcrystalline cellulose taken once daily for 28 days
Arm/Group | Mitoglitazone 90 mg | Mitoglitazone 220 mg | Pioglitazone 45 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
uIU/mL | 0.74 (4.664) | -9.77 (4.785) | -12.24 (5.215) | -1.60 (4.552)

3. Secondary Outcome: Change From Baseline in FFAs
Description: Change from baseline in Free Fatty Acids (FFAs)following 28 days of active therapy, as part of a lipid profile assessment
Time Frame: After 28 days of active therapy
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Mitoglitazone 90 mg | Mitoglitazone 220 mg | Pioglitazone 45 mg | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
mmol/L | -0.05 (0.051) | -0.15 (0.052) | -0.19 (0.057) | -0.01 (0.050)

4. Secondary Outcome: Change From Baseline in Triglycerides
Description: Change compared to baseline in triglycerides following 28 days of active therapy, as part of a lipid profile assessment
Time Frame: 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
mmol/L | 0.12 (0.160) | -0.21 (0.164) | -0.49 (0.179) | 0.15 (0.156)

5. Secondary Outcome: Change From Baseline in HDL
Description: Change from baseline in HDL following 28 days of active therapy, as part of a lipid profile assessment
Time Frame: 28 days
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
mmol/L | 0.00 (0.034) | 0.11 (0.034) | 0.09 (0.038) | -0.03 (0.033)

6. Post Hoc Outcome: Change From Baseline in FPG
Description: Change from baseline in fasting plasma glucose (FPG) following 28 days of active therapy
Time Frame: 28 days
Population: All patients who were compliant during the treatment period and who had Day 8 and Day 43 fasting plasma glucose values. Compliance during the treatment period was determined by the sponsor through a manual review of pill counts, including a review of comments from the study sites.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
mmol/L | -0.20 (0.263) | -0.97 (0.270) | -1.38 (0.294) | -0.04 (0.257)

7. Post Hoc Outcome: Change From Baseline in Insulin
Description: Change from Baseline in insulin levels following 28 days of active therapy
Time Frame: 28 days
Population: All patients who were compliant during the treatment period and who had a Day 8 and Day 43 pre-dose laboratory assessments. Compliance during the treatment period was determined by the sponsor through a manual review of pill counts, including a review of comments from the study sites.
Measure: Least Squares Mean (Standard Error); unit: uIU/mL
Arm/Group | MSDC-0160 90 mg | MSDC-0160 220 mg | Pioglitazone | Placebo
Number analyzed (Participants) | 20 | 19 | 16 | 21
uIU/mL | -5.01 (1.820) | -2.91 (1.867) | -6.58 (2.034) | -0.70 (1.776)

ADVERSE EVENTS:
Arm/Group | MSDC-0160 90 mg | Placebo | Pioglitazone | MSDC-0160 220 mg
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 4/22 | 3/22 | 2/21 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSDC-0160 90 mg (N=22) | Placebo (N=22) | Pioglitazone (N=21) | MSDC-0160 220 mg (N=21)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Peripheral Oedema (General disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less